CLINICAL TRIAL: NCT06596616
Title: MR Image Quality and Liver Lesion Detection With Gadopiclenol: Comparison With Gadoxetate Disodium
Brief Title: Gadopiclenol vs Gadoxetate MRI for Liver Lesions
Status: Enrolling by invitation | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Sara Lewis, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 23-1475
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Liver Lesion
MeSH Terms: interventions — X-Rays; gadopiclenol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Liver: Patients who have had clinically indicated MRI scans for liver lesions.
  Interventions: Other: Radiology; Other: Gadopiclenol

INTERVENTIONS:
Other: Radiology — Radiology - MRI Scans
Other: Gadopiclenol — Gadopiclenol is a new macrocyclic gadolinium-based contrast agent (GBCA)

SUMMARY:
The overall purpose of this study is to establish noninferiority of gadopiclenol MRI compared to gadoxetate MRI in terms of image quality and lesion detection/conspicuity in patients undergoing clinically indicated liver MRI in a prospective study. The research will be utilizing MRI; with enrollment goal of 75 subjects over the course of two years.

DETAILED DESCRIPTION:
Gadopiclenol is a new macrocyclic gadolinium-based contrast agent (GBCA) which has higher relaxivity than other GBCAs with a potential use of lower dose and comparable pharmacokinetics to other agents in preclinical studies. In a rodent model of liver metastasis, gadopiclenol showed strong enhancement with comparable pharmacokinetics to other extracellular GBCAs (EC-GBCAs). It was found to have a potential of either improving lesion conspicuity or providing similar accuracy in lesion detection with a reduced Gadolinium (Gd) dose. In a rat brain tumor model, half dose (0.05 mmol/kg) of gadopiclenol yielded comparable contrast-to-noise ratio (CNR) and morphological characterization of brain tumors compared to other EC-GBCAs. There are also a few clinical studies in which no safety concern was raised with the use of gadopiclenol. No dose adjustment for children or patients with renal impairment was found to be required. There is no study in the literature assessing the enhancement properties of gadopiclenol in abdominal imaging and comparing it with a hepatobiliary agent for image quality and lesion detection/conspicuity in the liver. For this study, it is hypothesized that dynamic imaging using Gadopiclenol is noninferior to gadoxetate MRI in terms of image quality and lesion detection/conspicuity.

ELIGIBILITY:
Inclusion criteria:

• Adult patients of both genders and all ethnic groups with clinical indication of MRI for chronic liver disease and/or focal lesion and/or tumor treatment follow-up.

Exclusion criteria:

* Acute renal insufficiency.
* Severe chronic renal insufficiency (GFR <30 mL/min/1.73 m2).
* Age <18y.
* Unable or unwilling to give informed consent.
* Contraindications for MRI (such as pacemakers, infusion pumps, pregnancy, allergy or previous adverse reactions to gadolinium contrast agents, severe claustrophobia).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with undergoing MRI for management of chronic liver disease, liver lesions, and/or tumor treatment follow up
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Lesion Detection | End of study, at 6 months
  Lesion detection (for any enhancing lesions including benign and malignant lesions, excluding cysts and completely necrotic treated malignant lesions) will be evaluated both for gadopiclenol-enhanced study (including unenhanced sequences from index MRI) and gadoxetate-enhanced MRI (the reference standard method): will be classified for each post- contrast phase as 0: no visible enhancing lesion, 1: visible enhancing lesion.

SECONDARY OUTCOMES:
Liver lesion conspicuity | End of study, at 6 months
  Liver lesion conspicuity (detected on full protocol clinical MRI scan) will be assessed for each postcontrast phase using the following scores: 0, not seen; 1: barely conspicuous; 2: fairly well seen; 3: moderately well seen; 4: well seen; and 5: very well seen. Each lesion will be delineated on Couinaud segmental maps.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lewis, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- BMEII, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Not within the scope the study